CLINICAL TRIAL: NCT06430879
Title: POWER-UP Trial (Performance Output With Haptics - Evaluating Athlete Response and Unrealized Potential)
Brief Title: Performance Output With Haptics - Evaluating Athlete Response and Unrealized Potential
Acronym: POWER-UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SuperPatch Limited LLC (Industry)
Collaborators: University of Arizona (Other); Clarity Science LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: POWER-UP 001
Record Dates: First submitted 2024-05-10; First posted 2024-05-28 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Muscle Strength; Muscle Weakness
Keywords: muscle; quadriceps; hamstrings; college athletes; elite athletes; haptic technology; vibrotactile trigger technology; VTT; neuromuscular changes
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo controlled, crossover trial with functional measurements
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active/Treatment (Active Comparator): Data will be collected for athletes prior to first use of patch and then 2-3 days later with the active patch (VICTORY PATCH). Follow-up functional measurements will also be taken at 7 and 9-10 days after baseline with second crossover patch use 9-10 days post-baseline.
  Interventions: Device: VICTORY PATCH
- Non-Active/Control (Sham Comparator): Data will be collected for athletes prior to first use of patch and then 2-3 days later with the inactive patch. Follow-up functional measurements will also be taken at 7 and 9-10 days after baseline with second crossover patch use 9-10 days post-baseline.
  Interventions: Device: Sham Patch without VTT
- Crossover (Other): Data will be collected for athletes prior to first use of patch and then 2-3 days later with the active or inactive patch. Follow-up functional measurements will also be taken at 7 and 9-10 days after baseline with second crossover patch use 9-10 days post-baseline.
  Interventions: Device: VICTORY PATCH; Device: Sham Patch without VTT

INTERVENTIONS:
Device: VICTORY PATCH — Drug- free, non-invasive patch (VICTORY Patch) with haptic vibrotactile trigger technology (VTT)
  Other Names: Haptic Vibrotactile Trigger Technology; VTT
  Arms: Active/Treatment; Crossover
Device: Sham Patch without VTT — Sham Patch without haptic vibrotactile trigger technology (VTT)
  Other Names: Sham Comparator
  Arms: Crossover; Non-Active/Control

SUMMARY:
This minimal risk, randomized, double-blind, placebo controlled Institutional Review Board (IRB)-approved observational study with functional measurements, will evaluate athletic performance after use of a drug- free, non-invasive patch (VICTORY Patch; The Super Patch Company Inc.); using KangaTech, Catapult and Force Plates along with crossover control of trials within the same subject group not receiving an 'active' patch.

DETAILED DESCRIPTION:
Emerging technologies that use haptic (skin pressure) technology have been studied and have shown positive improvements in stress levels, balance, sleep, and pain. The VICTORY patch (SuperPatch Company, Toronto, Canada) that also incorporates this technology has shown anecdotal promise to improve athlete performance. With the tools currently in use at the University of Arizona, team coaches and physicians can measure the true impact of neuromuscular changes suggested by the VICTORY patch. This study will measure quadriceps and hamstring strength in isolation as well as peak output in jumping and speed testing within in season training programs with and without VICTORY patch use. When combined with new methods of assessing individual muscle strength (KangaTech) and Force plate as well as Catapult measurements of compound movements of the investigational muscles, the investigators can evaluate the true performance and changes in football athletes with the SuperPatch technology.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 to 30, inclusive
2. Able to provide written informed consent
3. Have received a VICTORY Patch if in treatment group.
4. Is an athlete on a University of Arizona Varsity Athletic Team
5. Agree to having physical activity objectively measured for physical activity, as well as attendance, and participation in intervention.
6. Agree to place an adhesive patch on their skin, as instructed, based on selection group.

Exclusion Criteria:

1. Use of drugs of abuse (illicit or prescription)
2. Have an implanted device, or wears, or adheres any electrical device to the body during the study, other than a hearing aid.
3. Any current medical or musculoskeletal injury that would prohibit athletic participation
4. Any significant injuries in the last month prior to the intervention that may impact tested performance measures.
5. New injuries that occur during the course of study testing that may impact performance measures.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Changes in subject performance and strength and intensity/interference scores among and between the treated group and the control group for the athlete. | 10 days
  Evaluation of change in quadriceps and hamstring function via KangaTech measurements (mm/Kg)
Changes in subject performance and strength and intensity/interference scores among and between the treated group and the control group for the athlete. | 10 days
  Evaluation of change in max power of the Ground Reaction Force (GRF) in quadriceps and hamstring function measured by the Vald force plate (F = m * a ; 1 m/s2).
Changes in subject performance and strength and intensity/interference scores among and between the treated group and the control group for the athlete. | 10 days
  Evaluation of of Catapult Global Positioning System (GPS) and change in quadriceps and hamstring function to capture maximum acceleration and maximum speed (meters per second (m/s)) during their field workout.
Changes in subject performance and strength and intensity/interference scores among and between the treated group and the control group for the athlete. | 10 days
  Evaluation of change in subject response to The Borg Rating of Perceived Exertion (RPE) (scale= 1- 10)
Changes in performance based on patch location or playing position with the VICTORY Patch treatment. | 10 days
  Evaluation of performance (overall scores) based on concentration of patch placement among study subjects on either dominant medial forearm or dominant side, or mid-anterior thigh.

SECONDARY OUTCOMES:
Identification of subject phenotype(s) that will have the optimal response to treatment with the VICTORY Patch, as well as athletes having the least positive response. | 10 days
  Evaluation of predictive baseline metrics of playing position and predictive modeling will be used to identify subject phenotype(s) with an optimal, and a least positive, response. The data used as inputs to construct the predictive models will be a collection of the survey results collected from patients at day 0. Optimal and least positive responses will be defined based on changes in performance and other functional measurement scores, and changes in concomitant medications used, in the treatment group between survey dates.

OTHER OUTCOMES:
Any side effects reported by patients with be documented in athletic training electronic medical record and assessed by team physician and PI | 10 days
  Evaluation of reported side effects during study period based on self-report by subject or reported by clinician investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sakr, DO, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided